CLINICAL TRIAL: NCT05836129
Title: Effects of Transcendental Meditation on Rural Women of Lebanon
Brief Title: Lowering Stress Levels of Women in Lebanon
Acronym: TML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Responsible Party: Principal Investigator, Marie Loiselle, Director of Evaluation, Assistant Professor, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 30-62050-3816
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Stress; Resilience; Self Efficacy; Happiness
Keywords: Transcendental Meditation; Rural women in Lebanon
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The statistician will not be aware of which arm the participants are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TM Group (Experimental): The intervention used for this group is instruction in the Transcendental Meditation practice. It is a four day course of instruction with 1.5 hours of instruction over four consecutive days, followed by an additional 1.5 hours of instruction ten days later.
  Interventions: Behavioral: Transcendental Meditation (TM) practice
- Active Control Group (Active Comparator): This group will be offered an online stress reduction course consisting of two 20-60 minute classes for the first month of the trial.
  Interventions: Other: Stress reduction class (online)

INTERVENTIONS:
Behavioral: Transcendental Meditation (TM) practice — See previous description
  Arms: TM Group
Other: Stress reduction class (online) — See previous description
  Arms: Active Control Group

SUMMARY:
The goal of this clinical trial is to compare the experiences of women who learn the TM technique to those who do not. The main questions it aims to answer are:

1. Do women in rural Lebanon who practice the TM technique experience lower stress levels compared to those who do not.
2. Do women in rural Lebanon who practice the TM technique experience increased happiness, self-efficacy, and resilience levels compared to those who do not.

Participants will:

* complete baseline surveys
* be divided into experimental and active-control groups
* those in the experimental group will learn the TM technique, the control group will be offered an online didactic course on stress reduction
* both groups will complete post-test surveys at the end of 1 and 3 months

  * Researchers will compare experimental and control groups to see if the intervention effects stress levels.

DETAILED DESCRIPTION:
Methods: We will measure the effects of TM on 62+ women of the Chouf region of Lebanon using the following measures: Perceived Stress Scale, Connor-Davidson Resiliency Scale, New General Self-Efficacy Scale, and the Arabic Scale of Happiness. This is a randomized controlled trial with an experimental group and an active wait-list control group.

Measurements will be taken at baseline (pre-test) and at 1 and 3 months post-test.

ELIGIBILITY:
Inclusion Criteria: Females living in the Chouf region of Lebanon between the ages of 18-95.

-

Exclusion Criteria: Anyone: not female, under 18 or over 95, not in sound mental condition.

-

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Those who present as females.
Enrollment: 109 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 1 and 3-months on the Perceived Stress Scale(PSS-10) | Change = (week 12-baseline)
  The PSS measures the degree to which situations in one's life are appraised as stressful. Possible scores range from 0=never to 4=very often
Change from baseline to 1 and 3-months on the Connor-Davidson Resilience Scale (CDRS-10) | Change = (week 12-baseline)
  The CDRS-10 measures how well one is equipped to bounce back after stressful events, tragedy, or trauma
Change from baseline to 1 and 3-months on the Arabic Scale of Happiness (ASH-20) | Change = (week 12-baseline)
  The ASH-20 seeks to conduct a global, subjective assessment of whether a person is happy or unhappy
Change from baseline to 1 and 3-months on the New General Self-Efficacy Scale (NGSE-8) | Change = (week 12-baseline)
  The New General Self-Efficacy Scale assesses how much people believe they can achieve their goals, despite difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Fakhreddine, BA, Study Director — Chouf Development Council and the Ladies Foundation for Pure Knowledge
Locations (1):
- TM Home of Pure Knowledge Center, Beirut, Lebanon